CLINICAL TRIAL: NCT02207465
Title: A Phase I Dual Dose Escalation Study of Radiation and Nab-Paclitaxel in Patients With Unresectable and Borderline Resectable Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 32213
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced Unresectable Pancreatic Cancer Treated With Chemoradiotherapy; Borderline Resectable Pancreatic Cancer Treated With Chemoradiotherapy
MeSH Terms: interventions — Radiotherapy; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Subtrial 1-Arm A (Dose Level 1 of Abraxane) (Experimental): Determine if it is safe or not (via occurrence of dose limiting toxicities) for patients to receive both Abraxane and radiation therapy.
  Interventions: Radiation: Radiotherapy; Drug: Abraxane
- Subtrial 1-Arm B (Dose Level 2 of Abraxane: 3+4 enrollment) (Experimental): Determine the maximum dose of Abraxane that is allowable and safe for patients receiving both Abraxane and radiation therapy.
  Interventions: Radiation: Radiotherapy; Drug: Abraxane
- Subtrial 2- Abraxane 125mg; Borderline get 55cGY, unresectable get 57.5cGY until next escalation (Experimental)
  Interventions: Radiation: Radiotherapy; Drug: Abraxane

INTERVENTIONS:
Radiation: Radiotherapy
Drug: Abraxane — Dose varies within subtrial 1 to determine maximum dose. All patients in subtrial 2 receive 125mg Abraxane
  Other Names: nab-paclitaxel

SUMMARY:
The investigators hypothesize that intensification of local therapy will lead to improvements in local control and survival in patients with unresectable and borderline resectable pancreatic cancer. We propose to do this by combining nab-paclitaxel concurrently with dose-escalated radiation therapy. In the first part of this phase I study (sub-trial 1), the nab-paclitaxel dose will be escalated while the radiation dose is held constant at a standardly accepted level. The use of this novel chemoradiotherapy regimen will take advantage of nab-paclitaxel's specific anti-tumor and anti-stromal properties, which may enhance the efficacy of radiation therapy, and thereby improve local control. After the MTD of nab-paclitaxel had been determined, a second arm in sub-trial 1 will evaluate the addition of paricalcitol to nab-paclitaxel concurrently with dose-escalated radiation therapy. In addition, after the MTD of the nab-paclitaxel is reached in sub-trial 1 arm A, in the second part of this study (sub-trial 2), we will administer nab-paclitaxel at the determined MTD concurrently with escalated doses of radiation. We will utilize IMRT or protons to safely deliver high doses of radiation while maximally sparing surrounding normal tissue. Patients will also preferentially have 2-3 fiducial markers placed in or around the tumor for daily localization. Chemotherapy before and/or after chemoradiotherapy may be given as per standard of care. Correlative tissue and serum biomarkers are an important, but optional, part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed adenocarcinoma of the pancreas.
* Unresectable disease or borderline resectable disease assessed by a multidisciplinary panel of pancreas surgeon, medical and radiation oncologist, and a radiologist. Criteria defining unresectable and borderline resectable patients will be based on the NCCN Guidelines (v 1.2014):

Unresectable

* Greater than 180 degrees of SMA encasement
* Any celiac abutment
* Unreconstructible SMV/portal occlusion
* Aortic invasion or encasement
* Nodal metastases beyond the field of resection Borderline resectable
* Venous involvement of the SMV/portal vein demonstrating tumor abutment with impingement and narrowing of the lumen
* Encasement of the SMV/portal vein but without encasement of the nearby arteries
* Short-segment venous occlusion resulting from either tumor thrombus or encasement with suitable proximal and distal vessel for reconstruction/grafting.
* Gastroduodenal artery encasement up to the hepatic artery with either short segment encasement or direct abutment of the hepatic artery, without extension to celiac axis
* Tumor abutment to SMA but not to exceed greater than 180 degrees of circumferential vessel wall
* Age > 18 years.
* ECOG performance status of ≤ 1.
* Adequate organ function defined as follows: absolute neutrophil count of ≥ 1500/mm3, platelets ≥ 100,000/mm3, serum creatinine ≤ 2 mg/dl, total bilirubin ≤ 3, (with relief of biliary obstruction if present (PTC tube or endobiliary stent) and AST < 5 times the upper limit of normal.
* Patients of reproductive potential must agree to use an effective contraceptive method during participation in this trial and for 6 months after the trial.
* Patients must be able to provide written informed consent.

Exclusion Criteria:

* Distant metastatic disease.
* Prior history of abdominal radiation therapy.
* Prior systemic therapy for pancreatic cancer.
* Prior or simultaneous malignancy within the past 2 years (other than cutaneous squamous or basal cell carcinoma, melanoma in situ, thyroid carcinoma, or low-risk prostate cancer). In-situ carcinoma is allowed.
* Serious uncontrolled concomitant systemic disorders or psychiatric condition that would interfere with the safe delivery of protocol therapy.
* Treatment with an investigational anti-cancer agent within 4 weeks prior to enrollment into the study.
* Pregnant women, women planning to become pregnant and women that are nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2014-07; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Edgar Ben-Josef, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (2):
- United States (2):
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania